CLINICAL TRIAL: NCT04056923
Title: Three-dimensionally Printed Navigational Template for Localizing Small Pulmonary Nodules
Brief Title: 3D Printing for Nodule Localization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wen-zhao ZHONG (Unknown)
Collaborators: Zhuhai Seine Technology Co., Ltd, Zhuhai city, China (Unknown)
Responsible Party: Sponsor-Investigator, Wen-zhao ZHONG, M.D., Ph.D., Chief physician, Guangdong Provincial People's Hospital
Organization: GuangdongPPH (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3D printing navigation
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Pulmonary Nodule, Solitary; Lung Cancer
Keywords: Pulmonary Nodules; Lung Neoplasms; Computed Tomography; Three-Dimensional Printing
MeSH Terms: conditions — Solitary Pulmonary Nodule; Lung Neoplasms; Multiple Pulmonary Nodules | interventions — Indocyanine Green; Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D-printed template-guided(3D-G) (Experimental): Intraoperative 3D-G methylene blue dye marking in the operating room
  Interventions: Procedure: 3D-printing guided; Drug: Methylene blue; Procedure: Intraoperative
- CT-guided(CT-G) (Active Comparator): Preoperative localization is performed by CT-G indocyanine green marking in the radiology department
  Interventions: Procedure: CT-guided; Drug: Indocyanine Green; Procedure: Preoperative

INTERVENTIONS:
Procedure: 3D-printing guided — 3D printed navigational template guided
  Arms: 3D-printed template-guided(3D-G)
Procedure: CT-guided — CT-guided
  Arms: CT-guided(CT-G)
Drug: Indocyanine Green — The results are shown by comparison of different colors.
  Arms: CT-guided(CT-G)
Drug: Methylene blue — The results are shown by comparison of different colors.
  Arms: 3D-printed template-guided(3D-G)
Procedure: Preoperative — Preoperative localization.
  Arms: CT-guided(CT-G)
Procedure: Intraoperative — Intraoperative localization.
  Arms: 3D-printed template-guided(3D-G)

SUMMARY:
Implementation of lung cancer screening using low-dose computed tomography has increased the rate of detection of small peripheral pulmonary nodules. However, it is hard to localize these nodules by palpation because of their small volume and long distance to the nearest pleural surface. To further clarify the confounding factors, we developed our own 3D printing localization procedure. In contrast to traditional CT-G percutaneous puncture localization, our procedure was performed in the operating room without CT scan evaluation.

DETAILED DESCRIPTION:
Pulmonary wedge resection is one of the most common types of operations performed by thoracic surgeons, especially given that more and more patients with ground glass nodules are being detected recently. One of the most significant current discussion concerning wedge resection is nodule localization. At present, a commonly used localization method is the CT-guided percutaneous lung puncture methylene blue staining marker localization, but this method has two main disadvantages: 1. the methylene blue dye is easy to spread, affecting the intraoperative judgment of nodule position by surgeon; 2. patients often suffer additional CT radiation. In recent years, the three-dimensional (3D) printing technique has been gradually applied to clinical therapy. However, 3D-printed template-guided (3D-G) localization required pre-evaluation by CT scanning. If deviation of more than 2 cm was found on the CT scan, the 3D-G method was regarded as a failure and traditional CT-G hookwire localization was used. To further clarify the confounding factors, the investigators developed their own 3D printing localization procedure. In contrast to traditional CT-G percutaneous puncture localization, the 3D printing localization procedure was performed in the operating room without CT scan evaluation.

ELIGIBILITY:
Inclusion Criteria:

* a maximum target lung nodule diameter ≤20 mm;
* a target nodule consolidation/tumor ratio (CTR) <0.25, or a minimum distance from the outer edge of the nodule to the nearest pleural surface >10 mm if the target nodule CTR was >0.25.

Exclusion Criteria:

* Inability to comply with research protocols or research procedures
* Any unstable systemic disease (including active infections, uncontrolled high blood pressure, unstable angina, angina pectoris that has started within the last 3 months, congestive heart failure (≥ New York Heart Association [NYHA] Level II ), cardiac infarction (6 months before enrollment), severe arrhythmia requiring medication, liver, kidney or metabolic disease
* Active bleeding; Inability to withstand lying flat; Inability to cooperate through breathing during puncture
* Pregnant or lactating women
* Other circumstances that the investigator believes are not suitable for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Localization distance | Day of surgery
  The distance of the two stain points from the tumor. The investigators use a sterile, standard ruler to measure the distance. Based on our previous experience with CT-G localization, a deviation of less than 2 cm was considered a successful localization.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No